CLINICAL TRIAL: NCT00522990
Title: A Phase I/IIa Open-label Study to Assess the Safety, Tolerability and Preliminary Efficacy of AT9283, a Small Molecule Inhibitor of Aurora Kinases, in Patients With Refractory Hematological Malignancies
Brief Title: Study to Assess the Safety of Escalating Doses of AT9283, in Patients With Leukemias
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recommended Phase II dose determined
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT9283/0002; 2006-0177
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic Myeloid Leukemia; Myelodysplastic Syndromes; Myelofibrosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Primary Myelofibrosis | interventions — 1-cyclopropyl-3-(3-(5-morpholin-4-ylmethyl-1H-benzoimidazol-2-yl)-1H-pyrazol-4-yl)urea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Refractory Hematological Malignancies
  Interventions: Drug: AT9283

INTERVENTIONS:
Drug: AT9283 — Three weekly intravenous administration of AT9283

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of AT9283 that can be given to patients who have ALL, AML, CML, high-risk myelodysplastic syndromes, or myelofibrosis with myeloid metaplasia. Researchers want to perform pharmacokinetic (PK) testing on blood to find out how quickly the study drug leaves the body and how the body breaks down the drug. The safety and effectiveness of this drug will also be studied.

DETAILED DESCRIPTION:
Dose escalation study of AT9283 administered to patients with refractory hematological malignancies. Study objectives include identification of MTD and dose limiting toxicities, preliminary assessment of efficacy and definition of pharmacokinetic profile

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent
2. Histological or cytological confirmation of one of the following:

   Relapsed or refractory AML or ALL; acute leukaemia in patients who are unsuitable for or refuse standard therapy

   CML in chronic phase, accelerated phase or blast crisis that is resistant or refractory to standard therapy

   High-risk MDS, defined as the presence of:

   i)Refractory anemia with excess blasts (RAEB, 5-19% bone marrow blasts)

   or

   ii)RAEB in transformation to AML (RAEBT with 20-30% bone marrow blasts)

   Advanced MMM defined by the presence of one or more of the following features:

   i)Hemoglobin < 10 gm/dL (100 g/L)

   ii)Platelet count < 100 x 109/L

   iii)White blood cell count < 4 x 109/L

   iv)Symptomatic splenomegaly or other disease-related symptoms inadequately controlled by conventional therapies
3. ECOG performance status 0, 1 or 2
4. Male or female, age 18 years or older
5. Negative pregnancy test or history of surgical sterility or evidence of post-menopausal status (post-menopausal status is defined as any of the following: natural menopause with menses >1 year ago; radiation induced oophorectomy with last menses >1 year ago; chemotherapy induced menopause with 1 year interval since last menses

Exclusion Criteria:

1. Inadequate liver function as demonstrated by serum bilirubin ≥1.5 times the upper limits of reference range (ULRR) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or alkaline phosphatase (ALP) ≥2.5 times the ULRR (or ≥5 times the ULRR in the presence of liver metastases)
2. Impaired renal function as demonstrated either by an isolated creatinine value of ≥1.5 times the ULRR OR creatinine clearance < 50 mL/min determined by Cockcroft-Gault formula. Note there is no requirement to determine a formal creatinine clearance if the patient's serum creatinine value is ≥1.5 times the ULRR.
3. Radiotherapy or chemotherapy within the 14 days prior to the first dose of AT9283 being administered (Day 1, dose level 1). Planned use of hydroxyurea other than as is permitted as described in section 11.9.
4. Receiving an investigational anti-cancer treatment concurrently or within 14 days prior to the start of AT9283 infusion (Day 1)
5. Unresolved CTCAE grade 2 or greater toxicity (other than stable toxicity) from previous anti-cancer therapy excluding alopecia
6. Any evidence of severe or uncontrolled systemic conditions (e.g., severe hepatic impairment) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol
7. Active, uncontrolled central nervous system disease
8. Ischemic heart disease or myocardial infarction or unstable cardiac disease within 3 months of study entry
9. Prior infection with human immunodeficiency virus (HIV), hepatitis B or C viruses - screening for viral infections is not required for entry to this study
10. Major surgery within 28 days prior to the start of AT9283 infusion (Day 1) - excluding skin biopsies and procedures for insertion of central venous access devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 30 days after completing therapy with AT9283

SECONDARY OUTCOMES:
Pharmacokinetic profile, Safety and tolerability of maximum tolerated dose, efficacy, pharmacodynamic effect, identify dose limiting toxicities | Within six months of initiating therapy with AT92823

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Foran J, Ravandi F, Wierda W, Garcia-Manero G, Verstovsek S, Kadia T, Burger J, Yule M, Langford G, Lyons J, Ayrton J, Lock V, Borthakur G, Cortes J, Kantarjian H. A phase I and pharmacodynamic study of AT9283, a small-molecule inhibitor of aurora kinases in patients with relapsed/refractory leukemia or myelofibrosis. Clin Lymphoma Myeloma Leuk. 2014 Jun;14(3):223-30. doi: 10.1016/j.clml.2013.11.001. Epub 2013 Nov 14. PMID 24355079
- See also: Publication of the Study Results — http://www.ncbi.nlm.nih.gov/pubmed/24355079